CLINICAL TRIAL: NCT03704883
Title: Behavior of Cyclists in Response to Pain: a Qualitative Study
Brief Title: Behavior of Cyclists in Response to Pain
Status: Completed | Type: Observational
Sponsor: Allina Health System (Other)
Responsible Party: Sponsor
Other Study IDs: CKML-1601
Record Dates: First submitted 2018-10-08; First posted 2018-10-15 (Actual); Last update posted 2018-10-15 (Actual); Status verified 2018-10

CONDITIONS: Pain; Sport Injury; Athletic Injuries
Keywords: Cycling; Endurance; Pain; Injury
MeSH Terms: conditions — Pain; Athletic Injuries; Wounds and Injuries

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A qualitative study, as a follow-up to an earlier study, that provides an opportunity to develop a deeper understanding of the injured cyclist's behavior related to seeking medical attention and endurance of pain. This study includes 10 club-level cyclists who have an injury and either have or have not sought medical attention.

ELIGIBILITY:
Inclusion Criteria:

* Have at least one year of cycling experience and will not compete in multi-sport events such as a triathlon.
* Have had an injury currently or in the recent past associated with biking and experiencing pain related to cycling injury(s).
* Must read and speak English.

Exclusion Criteria:

* Non-English speaking

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Club-level cyclists, recruited from a local bike shop, who have an injury and either have or have not sought medical attention.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2016-05-01 (Actual); Primary Completion 2018-09-01 (Actual); Study Completion 2018-09-01 (Actual)

PRIMARY OUTCOMES:
Self-reported experience of cycling-related pain | Up to 30 minutes
  Key themes elicited from semi-structured interviews with participants. Themes will involve experiences related to cyclists' experience of pain and behavior related to pain, specifically the decision surrounding if and how to seek medical attention.

CONTACTS AND LOCATIONS:
Overall Officials: Marie C Lesiz, DO, Principal Investigator — Allina Health
Locations (1):
- Abbott Northwestern Hospital, Minneapolis, Minnesota, United States